CLINICAL TRIAL: NCT00224224
Title: A Comparison of Primary Care and Traditional Internal Medicine Residents
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Other Study IDs: 9510000400 (Formerly 1095-071)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Breast Cancer Screening; Cervical Cancer Screening; Cholesterol Screening; Asthma Admission Rate; Diabetes Management
Keywords: Clinical performance; Continuity of care; Utilization of resources

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to identify objective differences between primary care and traditional medicine residents in clinical performance, continuity of care and utilization of resources. Specifically, this retrospective study will analyze the database collected by CLIMACS, the computer system at Cornell Internal Medicine Associates (CIMA). This system is used for clinical and administrative purposes; it manages and tracks patient's information and demographics, appointment booking, clinical diagnosis, prescriptions and medications, laboratory and radiology test, and consults. In our study, we will analyze a subset of the CLIMACS database from previous years.

DETAILED DESCRIPTION:
Three areas will be examined:

1. Clinical performance
2. Continuity of care
3. Utilization of resources

Clinical performance will be assessed using Health Plan Employer data and Information Set (HEDIS) performance standards. These standards were developed for the purposes of quality assessment, and in our study we will examine the following HEDIS standards:

1. Breast Cancer Screening- the proportion of women between the ages of 52 and 64 who have had a mammogram within a two year period.
2. Cervical Cancer Screening- the proportion of women between the ages of 21 and 64 who had a Pap test in the preceding 3 years.
3. Cholesterol Screening- the proportion of patients ages 20 to 39 and 40-59 who have had their cholesterol tested at least once in the past five years.
4. Asthma admission rate- the proportion of asthmatics admitted to the hospital for the care of asthma per year.
5. Diabetic Standards-

   1. Admission for cellulitis/ 1000 diabetics per year.
   2. Admission for diabetes/ 1000 diabetics per year.
   3. Inpatient days per 100 diabetics per year.
   4. Prevalence of ischemic heart disease.
   5. Prevalence of severe renal disease.
   6. Diabetics with >2 hemoglobin A1C drawn per year.

Continuity of Care will be assessed by 3 different indicators:

1. The proportion of visits that are made to the designated primary care provider of the number of visits made.
2. The proportion of missed appointments of the total number of appointments.
3. The proportion of walk in visits of the total number of appointments.

Resource utilization will be assessed by examining the following:

1. Number of lab test per year per patient.
2. Number of specialty consults per year per patient.
3. Hospital admission rates per patient per year.
4. Cost to medications. Confidentiality will be maintained throughout the study. In clinical practice access to CLIMACS is limited to the medical providers and administrators by individuals access codes. Furthermore, our study will remove specific identifiers to maintain the anonymity of both the patients and residents.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are followed as outpatients by a Cornell affiliated internist at the Cornell Internal Medicine Associates (CIMA).
2. Patients at New York Hospital who may or may not go on to be followed as outpatients at CIMA.

Exclusion Criteria:

Patients who elect not to participate in the study.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1995-01; Study Completion 2005-01

PRIMARY OUTCOMES:
To identify the differences between primary care and traditional medicine residents in clinical performance, continuity of care and utilization of resources.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Medical College, New York, New York, United States